CLINICAL TRIAL: NCT03670641
Title: Remission Through Early Monitored Insulin Therapy - Duration Month
Acronym: REMIT-DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sandra Sobel (Other)
Responsible Party: Sponsor-Investigator, Sandra Sobel, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO17110070
Record Dates: First submitted 2018-09-06; First posted 2018-09-13 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Insulin therapy; Continuous glucose monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Intervention Model Description: 10 participants will be recruited soon after diagnosis of type 2 diabetes and started on short term insulin therapy to achieve euglycemia with insulin doses guided by continuous glucose monitor algorithm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Insulin and CGM Intervention (Experimental): 10 individuals with newly diagnosed type 2 diabetes will be started on basal (glargine) bolus (lispro) insulin therapy for up to 4 weeks with titrations guided by continuous glucose monitor (Dexcom G6) to achieve euglycemia and then insulin stopped after 4 weeks with hopes of diabetes remission.
  Interventions: Drug: Glargine; Drug: Lispro; Device: Dexcom G6

INTERVENTIONS:
Drug: Glargine — Dexcom G6 CGM will be used to guide daily insulin glargine and lispro dose titrations in participants with newly diagnosed type 2 diabetes. After 4 weeks of CGM and insulin therapy, insulin will be discontinued and participant's labs monitored every 3 months to determine if diabetes remission achieved.
  Other Names: Lantus
Drug: Lispro — Dexcom G6 CGM will be used to guide daily insulin glargine and lispro dose titrations in participants with newly diagnosed type 2 diabetes. After 4 weeks of CGM and insulin therapy, insulin will be discontinued and participant's labs monitored every 3 months to determine if diabetes remission achieved.
  Other Names: Humalog
Device: Dexcom G6 — Dexcom G6 CGM will be used to guide daily insulin glargine and lispro dose titrations in participants with newly diagnosed type 2 diabetes. After 4 weeks of CGM and insulin therapy, insulin will be discontinued and participant's labs monitored every 3 months to determine if diabetes remission achieved.
  Other Names: CGM

SUMMARY:
REMIT-DM is a feasibility pilot study where participants will be recruited soon after their diagnosis of type 2 diabetes to be placed immediately on insulin therapy for maximum of four weeks with titrations of insulin guided by glucose levels and trends provided by a continuous glucose monitor (CGM), with the purpose of achieving diabetes remission.

DETAILED DESCRIPTION:
REMIT-DM is a feasibility pilot study that aims to show that previously published diabetes remission through early use and titration of short-term insulin therapy is possible and safe in the ambulatory diverse American population of patients with T2D, with continuous glucose level and trend information provided by CGM. We developed the algorithm based on published diabetes remission studies and include within the algorithm the CGM trend arrows to further refine insulin doses for both safety and efficacy purposes. Data captured by the CGM transmits automatically to the cloud and is accessible at any time of day by the multidisciplinary diabetes team, which includes the certified diabetes educator (CDE) and Endocrinologist. The CGM-guided insulin titration algorithm is designed to achieve euglycemia (defined as fasting CBG < 100 mg/dL, and 2 hour post-prandial CBG < 120 mg/dL) within 2 weeks of initiating insulin therapy, then to help maintain euglycemia for 2 weeks before discontinuing insulin entirely. Ten participants will undergo a maximum of 4 weeks of insulin therapy and will be assessed for remission afterwards to confirm enough recovery of beta cell function. (Complete remission is defined as fasting glycemia <100 mg/dL without use of pharmacological therapy.) Afterwards, we will implement American Diabetes Association (ADA) guidelines for standard glycemic management, as necessary. We will use the data collected during this feasibility study to sharpen the CGM-guided insulin titration algorithm for creation of a T2DM remission mobile application that could then be tested and studied in a larger sample size.

The feasibility study will also take into account clinically meaningful data points e.g. the number of phone calls between the patient and the diabetes team, the patient experience, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. A1C criteria - >7.0
3. Newly diagnosed with T2D within 4 years
4. Lifestyle controlled
5. Subject may be on up to 2 medications for diabetes.
6. Smart phone or home computer compatible with DEXCOM CLARITY software
7. English speaking
8. Assessed by endocrinologist and diabetes educator to be able to perform skills necessary for CGM use and insulin delivery

Exclusion Criteria:

1. Autoimmune Type 1 DM, defined as positive GAD65 or islet cell antibodies
2. Pregnant
3. Chronic Kidney Disease (CKD) Stage IV or greater
4. Mental and/or cognitive disorder (based on documented disorder and/or assessment of physician or educator)
5. No access to computer for downloading CGM
6. BMI <18.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra I Sobel, MD, Principal Investigator — University of Pittsburgh; David A Rometo, MD, Principal Investigator — University of Pittsburgh; Linda Siminerio, RN PhD, Principal Investigator — University of Pittsburgh; Shari Reynolds, Study Chair — University of Pittsburgh
Locations (1):
- UPMC Falk Diabetes Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified using Pitt+Me, an online community which notifies patients about research studies they may be interested.
Period: Overall Study
Arm/Group | Insulin and CGM Intervention
Started | 10
Completed | 7 (3 participants were lost to follow up by 12 months)
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Insulin and CGM Intervention
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline A1C and A1C Measured at 3 Month Intervals up to 12 Months
Description: Blood test drawn at baseline and after insulin and CGM-guided titration intervention at 3 month intervals to see if improvement in aggregate A1C value is achieved.
Time Frame: Every 3 months up to 1 year
Population: Individuals recruited had newly diagnosed type 2 diabetes, never on insulin therapy. They may have been on other anti-hyperglycemic agents. The reason why the number analyzed in one or more rows differs from the overall number analyzed is because two of the patients unfortunately did not get baseline A1C measurements. and starting at month 6, 3 participants were lost to follow up
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Insulin and CGM Intervention
Number analyzed (Participants) | 10
percentage of glycosylated hemoglobin
  Pre-intervention: number analyzed (Participants) | 8
  Pre-intervention | 9.00 (1.56)
  3 months: number analyzed (Participants) | 9
  3 months | 6.81 (0.52)
  6 months: number analyzed (Participants) | 7
  6 months | 7.13 (1.43)
  9 months: number analyzed (Participants) | 7
  9 months | 7.26 (1.41)
  12 months: number analyzed (Participants) | 7
  12 months | 6.88 (1.20)

2. Secondary Outcome: Number of Participants With A1C of <6.5% After CGM-guided Insulin Therapy Intervention
Description: See if A1C achieves threshold <6.5% with intensive daily titration of basal bolus insulin therapy, guided by the individual's continuous glucose monitoring value and trend arrow - all guided by our algorithm.
Time Frame: A1C measures every 3 months up to 1 year
Population: These were the same 10 participants that were recruited at the beginning of the study, individuals with type 2 diabetes never on insulin therapy. We had one lost to follow up at 3 months and then 3 lost to follow-up at the remaining 3 month marks until completion of the study 1 year later
Measure: Count of Participants; unit: Participants
Groups:
- # of Participants With A1C <6.5%: This outcome determined the total number of participants that achieved A1C <6.5% at each 3 month interval up until conclusion of study at 12 months
Arm/Group | # of Participants With A1C <6.5%
Number analyzed (Participants) | 10
Participants
  3 months: number analyzed (Participants) | 9
  3 months | 1
  6 months: number analyzed (Participants) | 7
  6 months | 2
  9 months: number analyzed (Participants) | 7
  9 months | 2
  12 months: number analyzed (Participants) | 7
  12 months | 4

3. Secondary Outcome: Number of Patients With Glucose Values <55 mg/dL During 4 Week of Insulin and CGM Intervention
Description: We wanted to ensure that during the course of the intensive CGM-guided insulin therapy, our algorithm would be able to avoid severe hypoglycemia, defined as a glucose reading of <55mg/dL in the study participants
Time Frame: 4 weeks
Population: All participants with newly diagnosed type 2 diabetes were placed on CGM monitoring and had individualized insulin therapy for 4 weeks, with the goal of achieving predetermined glycemic targets. We wanted to see if any of the participants experienced severe hypoglycemia during this insulin intervention phase.
Measure: Count of Participants; unit: Participants
Groups:
- # of Participants Who Had a Continuous Glucose Reading <55mg/dL During Insulin Intervention Week: This was to capture if any of the participants had severe hypoglycemia, defined as <55mg/dL, during the 4 week insulin intervention.
Arm/Group | # of Participants Who Had a Continuous Glucose Reading <55mg/dL During Insulin Intervention Week
Number analyzed (Participants) | 10
Participants | 4

4. Secondary Outcome: See if Diabetes Distress is Affected With Intervention Via Problem Areas In Diabetes (PAID) - 5 Questionnaire Scale
Description: Administer the PAID-5 scale, which is a measure of diabetes distress. The scale ranges from a minimum of 0 (not a problem) to a maximum score of 4 (serious problem). The sum of the five questions provides the participant's score with a score range of minimum score of 0 to a maximum score of 20. A total score of greater than or equal to 8 indicates possible diabetes related emotional distress, with a higher score indicating more significant distress. This will be given to participants to see if/how distress levels change via the intervention
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Insulin and CGM Intervention
Number analyzed (Participants) | 10
units on a scale
  Pre-intervention | 8.90 (3.66)
  Post-intervention | 7.62 (4.35)

5. Secondary Outcome: Percent Time Glucose Values Remain in Range While Wearing CGM During Insulin Intervention
Description: Use CGM-captured glucose values to determine how often a participant's glucose levels were in range (percent time in range)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of time in range
Arm/Group | Insulin and CGM Intervention
Number analyzed (Participants) | 10
percentage of time in range
  Pre-intervention | 46.3 (28.4)
  Post-intervention | 80.67 (10.7)

6. Secondary Outcome: Number of Participants Achieving Euglycemic Glucose Targets Within a 4 Week Period
Description: The design of the algorithm was to attempt to achieve glucose values in the normal glycemic range, as defined as fasting BG target 80-95 mg/dL, and 2 hour post prandial BG target 100-120 mg/dL, within 2 weeks of starting insulin and maintaining values until end of 4 week intervention. We wanted to see if our CGM-guided insulin algorithm could help participants achieve pre-defined euglycemic glucose targets in four week period
Time Frame: 4 weeks
Population: The 10 participants analyzed were the same 10 participants recruited at the beginning of the study with newly diagnosed diabetes, never before on insulin therapy, using our CGM-guided insulin algorithm to try to achieve euglycemia within 4 weeks of therapy
Measure: Count of Participants; unit: Participants
Groups:
- # of Participants Achieving Glucose Targets: In this secondary outcome, we wanted to quantify the number of participants able to achieve a pre-specified fasting glucose of <95mg/dL within the first two weeks of insulin therapy. We also wanted to quantify the number of participants able to achieve a pre-specified 2 hour post-prandial glucose target of <120mg/dL within the first two weeks of insulin therapy.
  secondary outcome goals was for participants to be able to achieve fasting glucose levels <95mg/dL within two weeks of the CGM-guided insulin intervention. We report the number of participants who were able to do so
  One participant didn't titrate the insulin dose, one participant was lost to follow up, and two did not achieve goal fasting glucose in the first two weeks of therapy
Arm/Group | # of Participants Achieving Glucose Targets
Number analyzed (Participants) | 10
Participants
  Fasting Glucose <95 mg/dL | 6
  2hr post prandial glucose <120 mg/dL | 8

ADVERSE EVENTS:
Time Frame: 1 year post enrollment
Arm/Group | Insulin and CGM Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin and CGM Intervention (N=10)
Hypoglycemia (Endocrine disorders) | 7 (60) — This is defined as events of continuous glucose monitor or self-monitored blood glucose measure <70mg/dL that did not result in neuroglycopenia or require the assistance of others to resolve and was transient.
Signal Loss with Continuous Glucose Monitor (CGM) (Endocrine disorders) | 6 (6) — This captures the number of participants who had signal loss with their CGM from greater than 4 hours

LIMITATIONS AND CAVEATS:
Statistical analyses beyond those reported here were not conducted due to low number of participants enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03670641/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03670641/ICF_001.pdf